CLINICAL TRIAL: NCT03124316
Title: Testing a Behavioural Approach to Improving Cancer Screening Rates Through Increased Use of Primary Care Feedback Reports
Brief Title: Testing a Behavioural Approach to Improving Cancer Screening Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Ontario Institute for Cancer Research (Other); Cancer Care Ontario (Other); Ottawa Hospital Research Institute (Other); Laval University (Other)
Responsible Party: Principal Investigator, Noah Ivers, MD PhD, Women's College Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2017-004-E
Record Dates: First submitted 2017-04-18; First posted 2017-04-21 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Early Detection of Cancer; Clinical Trial

STUDY DESIGN:
Intervention Model Description: We will test three components of reminders to family physicians that could be embedded independently, in combinations of two, and all together in a reminder email. Family physicians will be randomly allocated to one of 8 experimental conditions. Each experimental condition comprises a different combination of the behaviour change techniques featured in the redesigned email reminder.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization schedule will be generated by a statistician on study IDs. The allocation sequence is applied simultaneously to the full set of eligible family physicians so that each is assigned to one of eight experimental conditions. The assignment to study conditions will be concealed from investigators. The data collection system used for the 4 month outcome assessment will be standardized across all study conditions and conducted by personnel at CCO not already involved in the study trial. No un-blinding is planned or permitted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Email #1: FULLY TURNED OFF (No Intervention): No behavioural change techniques (BCTs) 'turned on' in the email. The email would contain only standardized content.
- Email #2: ANTICIPATED REGRET (Experimental): Anticipated regret content + standardized content
  Interventions: Behavioral: Anticipated regret
- Email #3: MATERIAL INCENTIVE (Experimental): Material incentive content + standardized content
  Interventions: Behavioral: Material incentive
- Email #4: PROBLEM SOLVING (Experimental): Problem solving content + standardized content
  Interventions: Behavioral: Problem solving
- Email #5: REGRET + INCENTIVE (Experimental): Anticipated regret content + Material incentive content + standardized content
  Interventions: Behavioral: Anticipated regret; Behavioral: Material incentive
- Email #6: REGRET + PROBLEM SOLVING (Experimental): Anticipated regret content + Problem solving content + standardized content
  Interventions: Behavioral: Anticipated regret; Behavioral: Problem solving
- Email #7: INCENTIVE + PROBLEM SOLVING (Experimental): Material incentive content + Problem solving content + standardized content
  Interventions: Behavioral: Material incentive; Behavioral: Problem solving
- Email #8: ALL BCTs (Experimental): Anticipated regret content + Material incentive content + Problem solving content + standardized content
  Interventions: Behavioral: Anticipated regret; Behavioral: Material incentive; Behavioral: Problem solving

INTERVENTIONS:
Behavioral: Anticipated regret — Induce awareness of future regret about the unwanted behaviour
  Arms: Email #2: ANTICIPATED REGRET; Email #5: REGRET + INCENTIVE; Email #6: REGRET + PROBLEM SOLVING; Email #8: ALL BCTs
Behavioral: Material incentive — Inform that valued objects will be delivered if and only if that has been progress in performing the desired behaviours
  Arms: Email #3: MATERIAL INCENTIVE; Email #5: REGRET + INCENTIVE; Email #7: INCENTIVE + PROBLEM SOLVING; Email #8: ALL BCTs
Behavioral: Problem solving — Analyze or prompt the person to factors that influence the behaviour and select strategies that help overcome barriers
  Arms: Email #4: PROBLEM SOLVING; Email #6: REGRET + PROBLEM SOLVING; Email #7: INCENTIVE + PROBLEM SOLVING; Email #8: ALL BCTs

SUMMARY:
Family doctors can play a critical role in successfully arranging cancer screening tests to occur, especially if they know which patients are due for these tests. However, they don't always interact with or take advantage of registry data to this end. For example, in Ontario, the Screening Activity Report provides exactly this information to family doctors, helping them identify their patients who are overdue for screening. Unfortunately, less than half of family doctors regularly use the Screening Activity Report even though they get monthly email reminders. One possible reason is that the reminders they receive are not designed to compel action. They are easy for family doctors to miss or dismiss. This study will compare multiple different ways of designing the reminders. The different versions of the email are tested in a 2^3 factorial trial testing three behaviour change techniques to see which ones will lead to more family physicians interacting with the Screening Activity Report and at increasing the number of patients that get all the appropriate screening tests for cervical, breast, and/or colon cancer.

DETAILED DESCRIPTION:
Screening is an important way to prevent cancer-related death, but many Ontarians do not receive guideline-recommended screening for cervical, breast, and colon cancer. Family physicians can play a critical role in successfully increasing screening rates. A recent evaluation by members of our team suggests that Screening Activity Report (SAR) use is associated with improved cancer screening, but there remains substantial room for improvement. For the SAR to reach its full potential to decrease cancer-related death by improving screening rates, family physicians must regularly access it and take the appropriate actions. Currently, family physicians receive monthly email reminders, which state that new data are available, but do not describe the benefits of the SAR for physicians or their patients. It is easy to imagine how a busy doctor would fail to act upon such emails, resulting in suboptimal use of the SAR and leading to avoidable delays in cancer screening, and management. Indeed, CCO data show that less than half of recipients attend to this email and <7% click through to the SAR. The objectives for this trial are to compare different versions of the reminders in a randomized trial to identify the features that most increase use of the SAR. This is a pragmatic, 2^3 factorial trial, comparing behaviour change techniques incorporated within email reminders to doctors increase their use of the SAR. Participants are those who are already sent monthly emails by CCO regarding the SAR. The trial will randomly assign participants to one of eight modified emails to determine which content is most effective at driving SAR-use over 4 months. With an expected sample size of over 5700 family physicians, we anticipate power to see differences of 3% across experimental conditions.

ELIGIBILITY:
Family physicians are eligible if they have signed up for the SAR and already receive reminder emails as part of their registration process for the SAR with CCO.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5525 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
SAR access | 4 months
  The primary outcome will be whether eligible family physicians access the SAR during the 4 months of the trial (Yes/No)

SECONDARY OUTCOMES:
SAR access rate | 4 months
  Number of times the SAR was accessed
Adherence to screening guidelines for breast, colon, and cervical cancer in patients of eligible PCPs | 4 months
  Proportion of patients meeting screening guidelines for breast, colon, and cervical cancer; and efforts made by participants to access the SAR-use

OTHER OUTCOMES:
Process Measures: contact made with Cancer Care Ontario | 4 months
  Number of calls to CCO contact centre regarding the SAR

CONTACTS AND LOCATIONS:
Overall Officials: Noah Ivers, MD, PhD, Principal Investigator — Women's College Hospital
Locations (1):
- Cancer Care Ontario, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vaisson G, Witteman HO, Bouck Z, Bravo CA, Desveaux L, Llovet D, Presseau J, Saragosa M, Taljaard M, Umar S, Grimshaw JM, Tinmouth J, Ivers NM. Testing Behavior Change Techniques to Encourage Primary Care Physicians to Access Cancer Screening Audit and Feedback Reports: Protocol for a Factorial Randomized Experiment of Email Content. JMIR Res Protoc. 2018 Feb 16;7(2):e11. doi: 10.2196/resprot.9090. PMID 29453190
- See also: CCO SAR website — https://www.cancercare.on.ca/pcs/primcare/sar/